CLINICAL TRIAL: NCT03192267
Title: Early Rheumatoid Arthritis Lung Disease Study
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0282-16-FB
Record Dates: First submitted 2017-03-31; First posted 2017-06-20 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: newly diagnosed rheumatoid arthritis; lung disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, and whole blood for RNA/DNA isolation will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- No treatment: No treatment

SUMMARY:
Extra-articular (outside of joints) disease occurs in approximately 50% of rheumatoid arthritis (RA) patients, with the lung being a common site of involvement. The goals of this study are to investigate and characterize lung disease and its prevalence in early RA participants. This will be done through pulmonary function and high resolution chest computed tomography (CT), questionnaires, and serum studies. Another goal is to find novel biomarkers, such anti-malondialdehyde-acetaldehyde (MAA) antibodies, as predictors of lung disease in RA participants.

DETAILED DESCRIPTION:
Extra-articular (outside of joints) disease occurs in approximately 50% of rheumatoid arthritis (RA) patients, with the lung being a common site of involvement. The purpose of this study is to characterize the prevalence and classification of lung disease in participants with newly diagnosed rheumatoid arthritis by prospectively gathering information on lung imaging and function, comorbidities and novel biomarkers, such as anti-malondialdehyde-acetaldehyde (MAA). Specifically, the study would determine whether (MAA) adduct antibody concentrations predict computed tomography (CT) changes consistent with RA-lung involvement and determine whether anti-MAA antibody concentrations predict pulmonary function abnormalities in forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), and diffusion lung capacity of carbon monoxide (DLCO). An additional goal is to develop a cohort of newly diagnosed RA patients who can be followed long-term through electronic medical record (EMR) surveys, and biobank samples.

ELIGIBILITY:
Inclusion Criteria:

* 19-90 years of age
* Able to give informed consent
* Diagnosis of RA by a Rheumatologist using 2010 American College of Rheumatology (ACR) criteria within the past 2 years

Exclusion Criteria:

* Inflammatory arthritis that does not meet 2010 American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA)
* Pregnant

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: While new onset RA is more likely to occur in young to middle age adults, investigators would also like to study those with more long standing disease. In particular, older RA participants with cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
High Resolution Computed Tomography Chest Scan Results | Baseline (Visit 1 only)
  A high resolution computed tomography (CT) chest scan will be done at visit 1 to evaluate the presence of lung disease.

SECONDARY OUTCOMES:
Anti-malondialdehyde acetaldehyde Antibody Concentrations as Abnormality Predictors in Forced Vital Capacity | Baseline and 1 year follow-up
  Forced vital capacity (FVC), the total amount of air expelled after a deep breath, will be measured (liters) at baseline and 1-year follow-up. These values will be correlated with anti-malondialdehyde acetaldehyde (anti-MAA) antibodies, a novel biomarker for rheumatoid arthritis (RA).
Anti-malondialdehyde acetaldehyde Antibody Concentrations as Abnormality Predictors in Forced Expiratory Volume | Baseline and 1 year follow-up
  Forced expiratory volume in 1 second (FEV1), the amount of air exhaled in a forced breath, will be measured (liters) at baseline and 1-year follow-up. These values will be correlated with anti-malondialdehyde acetaldehyde (anti-MAA) antibodies, a novel biomarker for rheumatoid arthritis (RA).
Anti-malondialdehyde acetaldehyde Antibody Concentrations as Abnormality Predictors in Diffusion Lung Capacity of Carbon Monoxide | Baseline and 1 year follow-up
  Diffusion lung capacity of carbon monoxide (DLCO), the efficiency of gas exchange in the lungs, will be measured (mL/min/mmHg) at baseline and 1-year follow-up. These values will be correlated with anti-malondialdehyde acetaldehyde (anti-MAA) antibodies, a novel biomarker for rheumatoid arthritis (RA).

CONTACTS AND LOCATIONS:
Overall Officials: Tina D Mahajan, MD, Study Chair — University of Nebraska; Bryant R England, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No